CLINICAL TRIAL: NCT07089147
Title: The Role of the Paris Questionnaire in the Assessment of Postpartum Coccydynia: Associations With Quality of Life and Functional Outcomes
Brief Title: Postpartum Coccydynia and the Paris Questionnaire
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/044
Record Dates: First submitted 2025-07-17; First posted 2025-07-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-07

CONDITIONS: Postpartum; Coccydynia
Keywords: postpartum; coccydynia; paris questionnaire
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- females in the postpartum period: The study will include females aged between 18 and 65 years who have not previously received any treatment for coccydynia and who are within a maximum of 2 years postpartum. The study does not involve any intervention. Only a questionnaire will be administered to the females.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Paris questionnaire, EuroQool (EQ-5D-3L) Questionnaire, Low Back Outcome Score

SUMMARY:
The aim of this study is to investigate the presence of coccydynia (tailbone pain) in women who have given birth and to examine the relationship between the Paris Questionnaire and other relevant assessment tools. The relationship between the Paris questionnaire, the Low Back Outcome Score, and Quality of Life will also be evaluated.

DETAILED DESCRIPTION:
Females aged between 18 and 65 years who have given birth will be included in the study. The postpartum duration of eligible participants will range from a minimum of 6 weeks to a maximum of 2 years. At the beginning of the survey, participants will be informed about the study and asked to provide their informed consent.

Sociodemographic and clinical data including age, height, body weight, educational level, income status, family type, smoking status, engagement in regular physical activity, presence of chronic diseases, and obstetric history (i.e., most recent mode of delivery, number of pregnancies, number of births) will be recorded. Following this, participants will be asked to complete the Paris Questionnaire, the General Quality of Life Scale, and the Low Back Outcome Score. The relationships among the relevant questionnaires will be analyzed, and the association of the Paris Questionnaire with the other scales will be interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age
* Having not received any previous treatment for coccydynia
* Having given birth within the last 2 years at most

Exclusion Criteria:

* Those who have undergone surgical intervention on their spine
* Those with a history of malignancy
* Those with rectal or gynecological diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Females who have not previously received any treatment for coccydynia, who are within a maximum of 2 years postpartum, and who voluntarily agree to participate in the study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Paris Questionnaire | baseline
  The Paris questionnaire assesses patients' pain in different positions and consists of five items.This questionnaire exclusively assesses functional aspects and has a maximum score of 10. An increase in the total score indicates greater pain intensity.

SECONDARY OUTCOMES:
EuroQool (EQ-5D-3L) | baseline
  The General Quality of Life Scale is a tool developed to assess health-related quality of life. It consists of two parts. The first part defines the health profile across five dimensions: mobility, self-care, social life, pain, and psychological status. Each dimension includes three statements reflecting the severity of problems (1 = slight problems, 2 = moderate problems, 3 = severe problems). The second part includes a visual analogue scale, similar to a thermometer, on which respondents rate their current health or pain status on a scale from 0 to 100
Low Back Outcome Score | baseline
  The Low Back Outcome Score is a questionnaire used to evaluate the functional status and outcomes in individuals with low back pain. The Low Back Outcome Score (LBOS) consists of 13 items, each with a different scoring system. Pain is assessed separately. While all other items are scored on a four-point scale, their contributions to the total score vary based on item weightings. Three distinct scoring categories can be identified: items scored on a 9-point scale (pain, employment, domestic and sports activities) can receive 0, 3, 6, or 9 points; items scored on a 6-point scale (rest, treatment or consultation, analgesia, and sexual life) can receive 0, 2, 4, or 6 points; and items scored on a 3-point scale (sleep, walking, sitting, traveling, dressing) can receive 0, 1, 2, or 3 points. The total score is calculated by summing the points of all items and ranges from 0 to 75. Lower scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Akkoyun Sert, PhD, Study Director — KTO Karatay University
Locations (1):
- Kto Karatay University, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Peyton FW. Coccygodynia in women. Indiana Med. 1988 Aug;81(8):697-8. No abstract available. PMID 3171154
- [Result] Maigne JY, Rusakiewicz F, Diouf M. Postpartum coccydynia: a case series study of 57 women. Eur J Phys Rehabil Med. 2012 Sep;48(3):387-92. Epub 2012 Jul 23. PMID 22820826